CLINICAL TRIAL: NCT00969930
Title: Genetic Association Study Between Single Nucleotide Polymorphisms (SNPs) and Cognitive Performance in Young Bipolar Type I Patients: LICAVALGENE
Acronym: Licavalgene
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Responsible Party: Ricardo Alberto Moreno, Institute of Psychiatry, Mood Disorders Unit, School of Medicine, University of Sao Paulo
Other Study IDs: LICAVALGENE 2009
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2009-09

CONDITIONS: Bipolar
Keywords: COMT; ApoE; BDNF; executive function; bipolar; cognition; Cognitive deficits and Bipolar disease type I
MeSH Terms: conditions — Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- healthy controls
- BD type I patients

SUMMARY:
This is a genetic association study of cognitive impairment in young bipolar disease type I patients without medications in mania, depression, hypomania or mixed states.

DETAILED DESCRIPTION:
Introduction:

Cognitive impairment in bipolar disease (BD) patients is common and recent data suggests that it may be an endophenotype of the disease as it differs individually, persists during periods of euthymia and co segregates in families of BD patients. Cognition is a complex trait and is therefore likely to be underpinned by many genes, each with a relatively small effect. Performance in each domain of the neuropsychological assessment can be statistically linked to the functional activity of particular protein and by extension to the genetic variants accounting for theses functional differences.

Methods:

80 patients with BD type I (SCID DSM-IV), age from 18 to 35 years old, currently on mania, depression, hypomania or mixed state after medication wash out will be submitted to complete neuropsychological evaluation and genotyped for COMT (val158met, rs165599, -287, rs737865), ApoE (epsilon 4) and BDNF (val66met)and 80 healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* BD type 1
* non euthymia
* 18-35 y.o.

Exclusion Criteria:

* pregnancy
* organic disease
* use of drugs
* schizophrenia
* mental retardation
* illiterate

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young bipolar disease patients in mania, depression, hypomania or mixed states without medication use over the past 15 days.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-03 (Actual); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Cognitive deficits in BD patients are associated with COMT, ApoE and BDNF polymorphisms | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Psychiatry, School of Medicine University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Soeira-de-Souza MG, Bio DS, Dias VV, Martins do Prado C, Campos RN, Costa LF, Moreno DH, Ojopi EB, Gattaz WF, Moreno RA. SHORT COMMUNICATION: Apolipoprotein E genotype and cognition in bipolar disorder. CNS Neurosci Ther. 2010 Oct;16(5):316-21. doi: 10.1111/j.1755-5949.2010.00153.x. PMID 20406267